CLINICAL TRIAL: NCT04288284
Title: Emergency Curative Resection of Colorectal Cancer, Do it With Caution. A Comparative Case Series
Brief Title: Emergency Curative Resection of Colorectal Cancer
Status: Completed | Type: Observational
Sponsor: University of Alexandria (Other)
Responsible Party: Principal Investigator, Mohamed El Messiry, Ass. Professor, University of Alexandria
Other Study IDs: 0302761
Record Dates: First submitted 2020-02-25; First posted 2020-02-28 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Colorectal Cancer; Oncologic Complications and Emergencies
Keywords: Complicated colorectal cancer; Curative resection; Surgical and oncologic outcomes
MeSH Terms: conditions — Colorectal Neoplasms; Emergencies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Surgical specimens after curative resection of colorectal cancer
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Emergency group: Patients presented to emergency by complicated colorectal cancer ( Obstruction, bleeding or perforation)
  Interventions: Procedure: Curative resection of colorectal cancer
- Elective group: Patients presented with uncomplicated colorectal cancer for resection treatment
  Interventions: Procedure: Curative resection of colorectal cancer

INTERVENTIONS:
Procedure: Curative resection of colorectal cancer

SUMMARY:
The feasibility and efficacy of emergency curative resection of complicated colorectal cancer is still controversial. This prospective study aim is to assess surgical and oncologic outcomes after emergency compared to elective curative resection of colorectal cancer

DETAILED DESCRIPTION:
60 consecutive patients presented with complicated colorectal cancer managed by emergency surgery were included and compared to another 155 consecutive patients admitted during the same period with uncomplicated colorectal cancer managed by elective surgery. Both groups were compared regarding curative resection rate, early postoperative mortality and morbidity, 3-years tumor recurrence and survival rates.

ELIGIBILITY:
Inclusion Criteria:

* All patients presented with Potentially operable colorectal cancer
* No clinical or radiological evidence of metastatic disease

Exclusion Criteria:

* Patients received preoperative chemoradiation
* Patients with clinical or radiological evidence of metastatic disease
* Patients with intraoperative evidence of metastatic disease
* Patients with intraoperative evidence of irresectable disease
* Patients with incomplete follow up

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study included 60 consecutive patients presented by complicated colorectal cancer treated by emergency surgery at Alexandria University hospital between January 2015 and January 2017 (Group I). Another 155 patients with uncomplicated colorectal cancer treated by elective surgery during the same period were included (Group II).
Sampling Method: Probability Sample
Enrollment: 215 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Adequate oncologic resection | histopathological assessment of surgical specimens within 2 weeks postoperative
  Negative resection margins + adequate lymphadenectomy ( Lymph Nodes retrieved > 12)
early postoperative mortality after curative resection of colorectal cancer | within 90 days after surgery
  early death due to cause related to surgery
early postoperative morbidity after curative resection of colorectal cancer | within 90 days after surgery
  surgery-related complications

SECONDARY OUTCOMES:
Tumor recurrence | By the end of the 3 years follow up period
  either local or distant
Disease free survival | By the end of the 3 years follow up period
  % of patients survived without recurrence
Overall survival | By the end of the 3 years follow up period
  % of all patients survived either with or without recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Elmessiry, MD, PhD, Principal Investigator — Ass. Professor of Surgery

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ghazi S, Berg E, Lindblom A, Lindforss U; Low-Risk Colorectal Cancer Study Group. Clinicopathological analysis of colorectal cancer: a comparison between emergency and elective surgical cases. World J Surg Oncol. 2013 Jun 11;11:133. doi: 10.1186/1477-7819-11-133. PMID 23758762
- [Background] Biondo S, Marti-Rague J, Kreisler E, Pares D, Martin A, Navarro M, Pareja L, Jaurrieta E. A prospective study of outcomes of emergency and elective surgeries for complicated colonic cancer. Am J Surg. 2005 Apr;189(4):377-83. doi: 10.1016/j.amjsurg.2005.01.009. PMID 15820446
- [Background] Kim J, Mittal R, Konyalian V, King J, Stamos MJ, Kumar RR. Outcome analysis of patients undergoing colorectal resection for emergent and elective indications. Am Surg. 2007 Oct;73(10):991-3. PMID 17983065